CLINICAL TRIAL: NCT01367977
Title: Head Circumference Growth in Children With Ehlers-Danlos Syndrome Who Develop Dysautonomia ("POTS" -- Postural Orthostatic Tachycardia Syndrome)Later in Life -- a Retrospective Analysis
Brief Title: Head Circumference Growth in Children With Ehlers-Danlos Syndrome Who Develop Dysautonomia Later in Life
Status: Completed | Type: Observational
Sponsor: Genetic Disease Investigators (Other)
Responsible Party: Sponsor
Other Study IDs: 61/3528
Record Dates: First submitted 2011-06-05; First posted 2011-06-07 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2015-04

CONDITIONS: Ehlers Danlos Syndrome; External Hydrocephalus; Dysautonomia; Postural Orthostatic Tachycardia Syndrome; Venous Insufficiency
Keywords: Ehlers Danlos Syndrome; External Communicating Hydrocephalus; Dysautonomia; Postural orthostatic tachycardia syndrome; Chronic cerebrospinal venous insufficiency
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Autonomic Nervous System Diseases; Postural Orthostatic Tachycardia Syndrome; Venous Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ehlers-Danlos patients: Patients with diagnosed or suspected Classic or Hypermobile Ehlers-Danlos Syndrome

SUMMARY:
It is known that 33-50% of Classic and Hypermobile Ehlers-Danlos Syndrome patients eventually develop dysautonomia, otherwise known as "POTS" (Postural Orthostatic Tachycardia Syndrome). Some of these patients develop dysautonomia as a result of a retroflexed odontoid, Chiari 1 Malformation or cranial settling and the resulting basilar impression. Many Ehlers-Danlos patients suffer with the same symptomology with no evidence of a cause according to MRI imaging.

It is the author's hypothesis that low-level External Communicating Hydrocephalus appears to be responsible for the constellation of autonomic and cranial nerve symptoms, and if present in the very young, an analysis of head circumference growth in the first 15 months of life should reflect abnormally rapid head growth, supporting this hypothesis.

DETAILED DESCRIPTION:
It is known that 33-50% of Classic and Hypermobile Ehlers-Danlos Syndrome patients eventually develop dysautonomia, otherwise known as "POTS" - Postural Orthostatic Tachycardia Syndrome. Some of these patients develop dysautonomia as a result of a retroflexed odontoid, Chiari 1 Malformation or cranial settling and the resulting basilar impression. However, many Ehlers-Danlos patients suffer with the same symptomology with no evidence of cause according to MRI imaging. It is the author's hypothesis that low-level External Communicating Hydrocephalus appears to be responsible for the constellation of autonomic and cranial nerve symptoms, and if present in the very young, an analysis of head circumference growth in the first 15 months of life should reflect abnormally rapid head growth, supporting the hypothesis.

The investigators will evaluate the head circumference of Ehlers-Danlos patients who display dysautonomia later in life. The head circumference analyzed will be from birth to approximately 15 months of age, as the sutures of the skull generally fuse between 16 and 18 months. Additionally, pediatricians do not usually measure head circumference routinely beyond this age.

In a small subset of Ehlers-Danlos patients who developed postural orthostatic tachycardia syndrome in their childhood or teen years, retrospective analysis of their head circumferences indicates such megalocephaly. On average, the children's heads were found to increase from approximately the 35th percentile to over the 90th percentile. Their weights and lengths did not increase in the same fashion, although some of the children remained in the higher percentages for their length.

A review of literature indicates that studies of children with megalocephaly (not necessarily having the diagnosis of Ehlers-Danlos) were considered to have a benign condition ("Benign External Communicating Hydrocephalus") because CT's at the age of 2 or 3 years appeared normal and neurological exams also appeared normal. However, studies have also shown that a large percentage of these children exhibited delayed motor development and some of them had delayed speech development.In some studies these children were treated with Diamox, and in other studies the children were merely observed.

It is the author's hypothesis that delayed motor development found in Ehlers-Danlos children is due at least in part to hydrocephalus, and not merely due to flexible joints, as previously surmised.

It is the author's contention that mild symptoms of irritability, headaches, sleep disorders, emotional "fits", and the later development of dysautonomia were never considered in these studies, yet are the likely symptoms of a low level of pressure that continued to be exerted on the brains of these children.

High pressure on the brain (even if subtle) could be evidence of congenital CCSVI (cerebrospinal venous insufficiency) or increased CSF (cerebral spinal fluid) production, or the poor drainage of cerebral spinal fluid, or both. Retrospective examination of skull expansion is a necessary step to ascertain these possibilities, allowing for early treatment and the hope of avoidance of the neurological symptoms, and often disabling effects of dysautonomia (and/or multiple sclerosis). It is the author's contention that "Benign External Hydrocephalus" is not a benign condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis, or suspected diagnosis of Classic or Hypermobile Ehlers-Danlos Syndrome and dysautonomia
* Must be able to present their head circumferences, weight and length for the first 15 months of their lives

Exclusion Criteria:

* Patients unable to present their head circumferences, weight and length for the first 15 months of their lives
* Patients with dysautonomia due to stroke of the brain stem

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Classic or Hypermobile Ehlers-Danlos Syndrome with dysautonomia, found through social media forums, internet advertising, local support groups, physicians working with this subset of patients.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Measurement of Head Circumference in Ehlers-Danlos patients (retrospectively), between the ages of birth to 15 months of age. | Retrospectively, between patients' birth to 15 months of age
  Measurements of head circumferences, weight and length of children (retrospectively), will be compared to "normals" as established by the U.S. Department of Health and Human Services, Centers for Disease Control and Prevention (CDC), 2008.

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Driscoll, O.D., Principal Investigator — Genetic Disease Investigators
Locations (1):
- POTS Care, Colleyville, Texas, United States

REFERENCES:
- [Background] Alvarez LA, Maytal J, Shinnar S. Idiopathic external hydrocephalus: natural history and relationship to benign familial macrocephaly. Pediatrics. 1986 Jun;77(6):901-7. PMID 3714384
- [Background] Hakim A. Hypermobile Ehlers-Danlos Syndrome. 2004 Oct 22 [updated 2024 Feb 22]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1279/ PMID 20301456
- [Background] Milhorat TH, Bolognese PA, Nishikawa M, McDonnell NB, Francomano CA. Syndrome of occipitoatlantoaxial hypermobility, cranial settling, and chiari malformation type I in patients with hereditary disorders of connective tissue. J Neurosurg Spine. 2007 Dec;7(6):601-9. doi: 10.3171/SPI-07/12/601. PMID 18074684
- [Background] Kumar R. External hydrocephalus in small children. Childs Nerv Syst. 2006 Oct;22(10):1237-41. doi: 10.1007/s00381-006-0047-1. Epub 2006 Mar 23. PMID 16555081